CLINICAL TRIAL: NCT00922519
Title: An Observational Pilot Study of 18F-Sodium Fluoride (Na18F) Whole Body PET Scans in Patients for Whom 99m Tc MDP Bone Scans Would Normally be Indicated.
Brief Title: Observational Pilot Study of 18F-Sodium Fluoride (Na18F) Whole Body Positron Emission Tomography (PET) Scans for Imaging Bone
Status: Terminated | Type: Observational
Why Stopped: Retirement of former Qualified Investigator and lack of resources to complete study.
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: DX-FLU-001; NCT01065922 (obsolete NCT alias)
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Bone Scan
Keywords: Positron Emission Tomography; Sodium 18F-Fluoride; 99mTc-MDP; Bone Scan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: 18F-Sodium Fluoride (Na18F)

INTERVENTIONS:
Other: 18F-Sodium Fluoride (Na18F) — 200-400 MBq/injection, up to 6 doses of Na18F will be permitted per patient as part of acceptable disease assessment.

SUMMARY:
This study is being done to provide an alternative to bone scanning with technetium-99m (99mTc) labelled diphosphonates, and to document the safety of {18F}-Sodium Fluoride (Na18F) as a Positron Emission Tomography (PET) imaging radiopharmaceutical. Since the current availability of 99mTc was severely reduced because of the Chalk River shut down, alternative approaches to done scanning are needed. PET imaging with Na18F is one alternative approach to providing this critical clinical service.

DETAILED DESCRIPTION:
18F-Sodium Fluoride (Na18F) PET imaging is a nuclear medicine procedure, and its principal radiopharmaceutical, Na18F, has been used for scanning the skeleton for the spread of cancer for more that 30 years, but has not been approved by Health Canada because less expensive alternate drugs have been available (99mTc diphosphonates). Given the sudden and drastic change in the availability of 99mTc, an acceptable alternative for 99mTc-diphosphonates is needed as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient for whom 99mTc-MDP bone scans would normally be indicated
* If female of child-bearing potential and outside the window of 10 days since the last menstrual period, a negative serum or urine pregnancy test is required.
* Age greater than or equal to 15 years
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in the study
* If an oncology patient, the patient should have a Karnofsky Performance Scale Score greater than or equal to 50

Exclusion Criteria:

* Nursing or pregnant females
* Ages less than 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients for whom 99mTc MDP bone scans would normally be indicated
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2009-06-18 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Establish the feasibility of using locally produced 18F-Sodium Fluoride for PET bone scans as a substitute for 99mTc MPD | 1 year

SECONDARY OUTCOMES:
Demonstrate the safety of 18F-Sodium Fluoride by documentation of adverse events. | 1 year

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Sunnybrook Health Services Centre, Toronto, Ontario